CLINICAL TRIAL: NCT06109597
Title: Risk Factors and Diagnostic Performance of Predictors as a Screening Technique for Gestational Diabetes Mellitus: A Retrospective Cross-Sectional Study.
Brief Title: Risk Factors and Diagnostic Performance of Predictors as a Screening Technique for Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, fatimah khobrani, Associate consultant family medicine, King Abdulaziz Medical City
Other Study IDs: fatimahkhobrani
Record Dates: First submitted 2023-10-15; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 75 g glucose tolerance test — Pregnant patient who visited obstetric clinic , who did 75 g glucose tolerance test

SUMMARY:
Background Gestational diabetes mellitus (GDM) is a condition that can have negative impacts on both mother and baby. Detecting GDM early is crucial, and fasting plasma glucose (FPG) has been suggested as a possible screening method. This retrospective cross-sectional study aims to investigate potential risk factors and complications associated with GDM. Additionally, it aims to establish the diagnostic performance of predictive factors as a screening method for GDM.

Methods Data were collected from the medical records of 247 pregnant women who visited high-risk pregnancy outpatient clinics at King Abdul-Aziz Medical City in Jeddah between 2021 and 2022. The study investigated potential risk factors and complications associated with gestational diabetes mellitus (GDM), including impaired fasting glucose/impaired glucose tolerance (IFG/IGT), family history of diabetes mellitus (DM), and medical conditions. Moreover, the study evaluated the diagnostic performance of potential predictors as screening techniques for gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
This study was a hospital-based retrospective cross-sectional study. The study was conducted at the clinic of King Abdul-Aziz Medical City, a tertiary care hospital in Jeddah, Saudi Arabia. Data were collected from the target population through the use of medical records.

Study Population For this study, the investigators looked at all pregnant patients who visited high-risk pregnancy outpatient clinics at King Abdul-Aziz Medical City in Jeddah from 2021 to 2022. Our focus was on singleton pregnant women who received prenatal care services in Obstetrics clinics at King Abdul-Aziz Medical City. However, to ensure accurate and valid results, the investigators excluded pregnant women with diabetes mellitus or autoimmune diseases. By examining this specific population of pregnant women, the investigators aimed to investigate potential risk factors and complications associated with high-risk pregnancies.

Sampling technique and size:

The sampling technique for this study is non-probability consecutive sampling, which will include all pregnant patients who visited high-risk pregnancy outpatient clinics at King Abdul-Aziz Medical City in Jeddah from 2021 to 2022. The study aims to collect data from all members of the target population instead of sampling from a larger population.

Data Collection Technique and Tool The data collection tool was developed and face-validated by two consultants in the field. The tool was designed to collect data from the medical records of the participants, including their fasting blood glucose (FBG) levels and oral glucose tolerance test (OGTT) results. The tool was also used to collect information about the participants' obstetric history, demographic characteristics, and medical conditions

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant women who received prenatal care services in Obstetrics clinics at king Abdul-Aziz medical city.

Exclusion Criteria:

* Pregnant known to have diabetes mellitus.
* Participant with Autoimmune disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant patients who attend high risk pregnancy outpatient's clinic at national guard hospital in Jeddah during 2021-2022.
  Dependent Variable:
  OGTT - Fasting Blood Glucose - Weight - Pregestational BMI
  Independent Variable(s):
  Age, Gender, Medication, Gestational age, Chronic diseases, Family history, Past gyne and medical history.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Complications associated with gestational diabetes mellitus | 1 year
  The study investigated potential risk factors and complications associated with gestational diabetes mellitus (GDM), including impaired fasting glucose/impaired glucose tolerance (IFG/IGT), family history of diabetes mellitus (DM), and medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah M Khobrani, Associate, Principal Investigator — KAMC
Locations (1):
- Fatimah Khobrani, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT06109597/Prot_SAP_000.pdf